CLINICAL TRIAL: NCT01151059
Title: A Phase II, Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of AGRIPPAL® S1 Surface Antigen, Inactivated, Influenza Vaccine, Formulation 2010-2011, When Administered to Non-elderly Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of One Dose of Inactivated Trivalent Flu Vaccine Administered to Non-elderly Adult and Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V71_19S
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Seasonal Influenza
Keywords: seasonal influenza; vaccine

ARMS (1):
- Group 1 (Other): No comparator is administered, only one IM single dose of trivalent subunit inactivated influenza vaccine is administered during the vaccination visit
  Interventions: Biological: Trivalent subunit inactivated flu vaccine, Formulation 2010-2011

INTERVENTIONS:
Biological: Trivalent subunit inactivated flu vaccine, Formulation 2010-2011 — This phase II is performed as a multicenter study site in non-elderly adult and elderly subjects. Enrolled subjects received one single IM dose of trivalent subunit inactivated flu vaccine during the vaccination visit, according to the study protocol (follow-up period: till day 22).

SUMMARY:
The present study will evaluate the safety and immunogenicity in healthy people (non-elderly adult and elderly subjects) after one intramuscular (IM) dose of trivalent subunit inactivated flu vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Males and females volunteers of 18 years of age or older, mentally competent, willing and able to give written informed consent prior to study entry
* Individuals able to complain with all the study requirements
* Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.

Exclusion Criteria:

* Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study
* Individuals with any serious chronic or acute disease (in the judgment of the investigator), including but not limited to: cancer, advanced congestive heart failure, chronic obstructive pulmonary disease (COPD), autoimmune diseases, acute or progressive hepatic and renal disease, severe neurological or psychiatric disorder and severe asthma
* Individuals with history of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study vaccine (e.g. to eggs/eggs product as well as ovalbumin, chicken protein, chicken feathers, influenza viral protein, kanamycin and neomycin sulphate)
* Individuals with known or suspected impairment/alteration of immune function resulting, for example, from: receipt of immunosuppressive therapy within the past 60 days and for the full length of the study, receipt of immunostimulants, receipt of parenteral immunoglobulin preparation, blood products and/or plasma derivates within the past 3 months and for the full length of the study and suspected or known human immunodeficiency virus (HIV) infection or HIV-related disease
* Individuals with known or suspected history of drug or alcohol abuse
* Female who are pregnant or nursing (breastfeeding) mothers or females of childbearing potential do not plan to use acceptable birth control measures for the whole duration of the study
* Individuals with history or any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study
* Individuals within the past 6 months, they have had any seasonal or pandemic laboratory confirmed influenza disease and received any seasonal or pandemic influenza vaccine
* Individuals with any acute or chronic infections requiring systemic antibiotic treatment or antiviral therapy within the last 7 days
* Individuals that have experienced fever (i.e., axillary temperature ≥ 38°C) within the last 3 days of intended study vaccination
* Individuals participating in any clinical trial with another investigational product 4 weeks prior to first study visit or intent to participate in another clinical study at any time during the conduct of this study
* Individuals who received any other vaccines within 4 weeks prior to enrollment in this study or who are planning to receive any vaccine within 4 weeks from the study vaccines
* Individuals who have ever received blood/blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 12 weeks and for the full length of the study
* Individuals who are part of study personnel or close family members conducting this study
* Individuals with a bleeding diathesis or conditions associated with prolonged bleeding time that in the investigator's opinion would interfere with the safety of the subject
* BMI > 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the antibody response to each influenza vaccine antigen at 21 days post-immunization in non-elderly adult and elderly subjects | 22 days, including the follow-up period

SECONDARY OUTCOMES:
To evaluate the safety of a single IM injection of trivalent subunit inactivated FLU vaccine in non-elderly adult and elderly subjects | 22 days, including the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (5):
- Italy (5):
  - Dipartimento di Medicina e Scienze dell'Invecchiamento, Università G. D'Annunzio, Via dei Vestini, Chieti
  - Dipartimento di Medicina Clinica e Sperimentale - Sezione di Igiene e Medicina Preventiva, Via Fossato di Mortara, 64/b, Ferrara
  - Dipartimento di Scienze della Salute Università di Genova Via Pastore, 1, Genova
  - Centro Satellite. ASL Lanciano - Vasto, sede legale Via S. Spaventa, 37, Lanciano
  - Vaccine and Immunotherapy Research Center Department of Infectious and Tropical Diseases San Raffaele Scientific Institute Via Stamira d'Ancona, 20, Milan